CLINICAL TRIAL: NCT04074512
Title: Copper Histidinate Treatment for Menkes Disease
Status: Available | Type: Expanded Access
Sponsor: Sentynl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CYP-001
Record Dates: First submitted 2019-08-27; First posted 2019-08-30 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-06

CONDITIONS: Menkes Disease
MeSH Terms: conditions — Menkes Kinky Hair Syndrome | interventions — copper bis(histidinate)

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: copper histidinate — copper histidinate for subcutaneous injection
  Other Names: CUTX-101

SUMMARY:
This expanded access protocol provides subcutaneous copper histidinate for Menkes disease patients under 6 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have been treated in protocol 09-CH-0059 or must be a newly diagnosed Menkes disease patient in the US.
2. Parent or legal guardian is willing and able to sign and date an informed consent form.
3. Male or female, aged 0 to <6 years of age.
4. Diagnosis of Menkes disease: A confirmed gene mutation in ATP7A is not required; however, the test must be at least pending prior to initiating therapy. For those patients whose molecular ATP7A gene mutation confirmation is pending, they should have serum copper <75 mcg/dL. If the mutation is subsequently not confirmed, the patient should discontinue treatment.
5. Ability to adhere to the prescribed subcutaneous copper histidinate injection regimen.
6. Willingness to adhere to all recommended visits and procedures.
7. Resident of the US.

Exclusion Criteria

1. Diagnosis of Wilson disease.
2. Any disease or condition that, in the opinion of the Investigator, has a high probability of precluding the subject from completing the study or where the subject cannot or will not appropriately comply with study requirements.
3. Receipt of concomitant medication or device not approved for any use (i.e. experimental) by FDA within 30 days prior to screening for this study, except for participation in protocol 09-CH-0059.
4. Patient/caregiver cannot or will not appropriately comply with protocol recommendations (e.g., site visits, renal monitoring).
5. Currently receiving any concomitant copper-containing medications.

Ages: 0 Years to 6 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California Davis Medical Center, Sacramento, California
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Memorial Healthcare Systems, Hollywood, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Emory University, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Maine Medical Center, Portland, Maine
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Shodair Children's Hospital, Helena, Montana
  - Duke University Hospital, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Monroe Carrell Jr. Children's Hospital at Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Health Care System, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- See also: Related Info — https://sentynl.com/